CLINICAL TRIAL: NCT03487770
Title: A Multicenter, Randomized, Double-blind, Flexible-dosed, Placebo-controlled, Parallel-group Clinical Trial Evaluating the Efficacy and Safety of Aripiprazole Oral Solution in Children and Adolescents With Autistic Disorder
Brief Title: Aripiprazole Oral Solution in the Treatment of Children and Adolescents With Autistic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-403-00106
Record Dates: First submitted 2018-03-27; First posted 2018-04-04 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-01

CONDITIONS: Autistic Disorder
Keywords: Autistic; Aripiprazole Oral Solution
MeSH Terms: conditions — Autistic Disorder | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole Oral Solution (Experimental): 1 mg/mL, 2 ~ 15 mg/day (2 ~ 15 mL/day), taken once daily for 8 weeks. Administrate about at the same time each day, either before or after meals;
  Interventions: Drug: Aripiprazole Oral Solution
- Placebo Oral Solution (Placebo Comparator): 2 ~ 15 mg/day (2 ~ 15 mL/day), taken once daily for 8 weeks. Administrate about at the same time each day, either before or after meals.
  Interventions: Drug: Placebo Oral Solution

INTERVENTIONS:
Drug: Aripiprazole Oral Solution — Aripiprazole 2~15 mg/day (2~15 mL/day)
  Other Names: Abilify; Aripiprazole
  Arms: Aripiprazole Oral Solution
Drug: Placebo Oral Solution — Placebo 2~15 mg/day (2~15 mL/day)
  Other Names: Placebo
  Arms: Placebo Oral Solution

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the efficacy, safety, tolerability and the steady-state plasma trough concentration of aripiprazole flexible-dosed in children and adolescents with a diagnosis of Autistic Disorder. Approximately 100 subjects will be randomly assigned at a 1:1 ratio to receive aripiprazole (2 to 15 mg) or placebo treatment for 8 weeks

DETAILED DESCRIPTION:
Screening Phase: up to 42 days (consisting of a Screening Visit (V1), a washout period and Interim Screening Visit (V1a) when applicable, and a Baseline Visit (V2). The Screening Phase will serve multiple purposes: to allow for appropriate washout of prohibited medications; to allow for review of screening data; to establish a pre-treatment baseline of key outcome measures.

Treatment Phase: The duration of the treatment is 8 weeks. The purpose of the treatment phase is to evaluate the efficacy, safety, tolerability and steady-state plasma trough concentration of aripiprazole in the treatment of serious behavioral problems in children and adolescents with a diagnosis of Autistic Disorder..

Safety Follow-up Phase: All subjects will be followed up for safety (adverse events) at Day 16 after the last medication via telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from a legally authorized guardianprior to the initiation of any protocol-required procedures.
2. The subject and/or the designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, in the opinion of the Investigator.
3. The patient meets current DSM-IV-TR diagnostic criteria for Autistic Disorder and also demonstrates behaviors such as tantrums, aggression, self-injurious behavior, or a combination of these problems. In addition, the Childhood Autism Rating Scale (CARS) score is ≥30.
4. The subject has a Clinical Global Impressions-Severity (CGI-S) score ≥ 4 AND an ABC-I subscale score ≥18 at screening (Visit 1 or Visit 1a) and baseline (V2).
5. Environmental factors can be consistent throughout the trial period.
6. The subject is a male or female child or adolescent 6 to 17 years of age (6 ≤ age ≤ 17) at Baseline (V2).

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the study.

   Note: WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea 12 consecutive months; or women on hormone replacement therapy with documented serum follicle stimulating hormone level ≥ 35 mIU/mL].
2. Women with a positive pregnancy test or who are pregnant or breastfeeding.
3. The subject has a current diagnosis of psychotic disorder such as bipolar disorder, schizophrenia, or depression.
4. The subject is currently diagnosed with another disorder on the autism spectrum, including Pervasive Developmental Disorder-Not Otherwise Specified, Asperger's Disorder, Rett's Disorder, Childhood Disintegrative Disorder or Fragile-X Syndrome.
5. The subject has a history of neuroleptic malignant syndrome.
6. The subject represents a significant risk of committing suicide based on history or routine psychiatric status examination.
7. The subject has had a seizure in the past year or the electroencephalograph examination is epileptiform discharge at screening.
8. The subject has a history of severe head trauma or stroke；
9. The subject has a history or current evidence of any unstable medical conditions (eg. history of congenital heart disease or arrhythmia, or cancer) that, in the judgment of the investigator would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial.
10. Non-pharmacological therapy (e.g., psychotherapy, behavior modification, and education training, etc.) could not be stable prior to screening and consistent throughout the study, and the subject who needs to use acupuncture and moxibustion, auditory integration, biofeedback and transcranial magnetic stimulation therapy as supplemental replacement therapy in 7 days prior to taking investigational product or during the course of the trial.
11. The subject is considered treatment resistant to antipsychotics medication, in the opinion of the Investigator, based on lack of therapeutic response to 2 different antipsychotics with reasonable doses after treatment of at least 3 weeks each.
12. The subjects considered treatment resistant to aripiprazole in the opinion of the investigator based on lack of therapeutic response to an adequate dose and duration of aripiprazole treatment.
13. The following laboratory test results, vital sign and Electrocardiograph (ECG) findings are exclusionary:

    * QTc > 450 msec (male), QTc > 470 msec (female)
    * Platelets (below the lower limit)
    * Hemoglobin (below the lower limit)
    * Neutrophils (below the lower limit)
    * AST (SGOT) or ALT (SGPT) (above the upper limit)
    * Creatinine (above the upper limit) In addition, subjects should be excluded if they have any other abnormal laboratory test result, vital sign result or ECG finding that in the investigator's judgment is clinically significant, in that it would impact the safety of the patient or the interpretation of the study results.
14. The subject weighs < 15 kg.
15. The subject has a known allergy or hypersensitivity to aripiprazole or other dihydrocarbostyrils (eg. carteolol, vesnarinone, and cilostazol).
16. The subject has participated in any clinical trials with an investigational agent within the past month.
17. Subjects who are likely to require prohibited concomitant therapy during the trial (refer to Section 7 Prohibited and Restricted Therapies).
18. Subjects who participated in a previous clinical trial of aripiprazole (with the exception of Investigator Sponsored Trials).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline to Week 8 (or endpoint) in the ABC-I score | Baseline and 8 weeks (or endpoint)
  The objective of the primary analysis is to compare the efficacy of aripiprazole flexible-dosed (2 ~ 15 mg/day) with placebo in reducing serious behavioral problems, specifically irritability, agitation and self-injurious behavior, in children and adolescents with a diagnosis of Autistic Disorder. The efficacy is assessed by assessed by change from baseline to endpoint on the Irritability Subscale of the ABC (ABC-I).

SECONDARY OUTCOMES:
Clinician-rated CGI-I score at Week 8 (or endpoint) | Baseline and 8 weeks (or endpoint)
  The efficacy is assessed by the clinician-rated CGI-I score at Week 8
Change in ABC subscale scores from Baseline to Week 8 (or endpoint) | Baseline and 8 weeks (or endpoint)
  The efficacy is assessed by changes from Baseline to Week 8 (or endpoint) in Social Withdrawal, Hyperactivity, Stereotypy and Inappropriate Speech Subscale scores of the ABC
Response Rate at Week 8 (or endpoint) (or endpoint) | Baseline and 8 weeks (or endpoint)
  The response is defined as a reduction ≥25% in ABC-I score compared to the baseline, and a CGI-I score of much improved or very much improved) at Week 8 (or endpoint).The efficacy is assessed by response rate at Week 8 (or endpoint).

CONTACTS AND LOCATIONS:
Overall Officials: Patyman Juma, Study Director — Otsuka Beijing Research Institute
Locations (1):
- 6th affiliated hospital, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No